CLINICAL TRIAL: NCT07336875
Title: Clinical Study of Novel CAR-ITNK Cells Targeting CD70 and CLL1 for Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: Clinical Study of Novel CAR-ITNK Cells Targeting CD70 and CLL1 for Refractory/Relapsed AML
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jia Wei, professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202512163
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: R/R AML
Keywords: CAR-ITNK; CD70&CLL1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Administer a single infusion of CAR-ITNK Cells targeting CD70 and CLL1 to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion, and conduct follow-up surveys at the required time points within three years post-infusion according to the visit schedule.
  Interventions: Biological: CAR-ITNK Cells targeting CD70 and CLL1

INTERVENTIONS:
Biological: CAR-ITNK Cells targeting CD70 and CLL1 — Administer a single infusion of CAR-ITNK Cells targeting CD70 and CLL1 to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of CAR-ITNK cells therapy targeting CD70 and CLL1 in participants with relapsed/refractory Acute Myeloid Leukemia. Participants will receive a single infusion of CAR-ITNK cell therapy targeting CD70 and CLL1 and complete follow-ups over the next three years.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a hematological malignancy disease originating from the bone marrow, typically presenting with acute onset, and patients may experience symptoms such as anemia, bleeding, and infections. The main treatment modalities currently include chemotherapy, targeted drug therapy, and hematopoietic stem cell transplantation. In addition to its low cure rate, AML has a high recurrence rate, is prone to developing resistance to chemotherapy drugs, and can easily lead to severe side effects, such as infections and bone marrow suppression. Therefore, there is an urgent need to find new therapeutic approaches for treating acute myeloid leukemia.

The research team at Guangdong Zhaotai Cell Biotechnology Co., Ltd. has independently developed and constructed a novel tandem CAR-ITNK cell targeting CD70 and CLL1. In vitro cytotoxicity assay data show that the activity of the tandem CAR-ITNK cells targeting both CD70 and CLL1 (CAR70C1-ITNK) in killing CD70- and CLL1-overexpressing cells is stronger than that of single-targeted CAR-ITNK cells against either CD70 or CLL1. In vivo xenograft mouse models using THP-1 cells demonstrate that the ability of CAR70C1-ITNK cells to kill THP-1 cells is superior to that of single-targeted CD70 CAR-ITNK cells. These experimental data indicate the potential value of the novel tandem CAR-ITNK cells targeting CD70 and CLL1 in clinically treating patients with refractory/relapsed acute myeloid leukemia.

This clinical trial proposes to use the novel tandem CAR-ITNK cells targeting CD70 and CLL1 as an interventional measure for subjects with refractory/relapsed acute myeloid leukemia. After treatment with these novel tandem CAR-ITNK cells, the safety and preliminary efficacy will be evaluated through various assessment methods, including clinical symptom evaluation, biomarker testing, laboratory tests, imaging assessments, adverse event monitoring, and follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their legal guardian voluntarily participates and has signed the informed consent form.

2. Age between 18 and 75 years old (inclusive), with no gender restrictions. 3. Diagnosed as having refractory/relapsed acute myeloid leukemia, meeting one of the following criteria:

1. . Reappearance of leukemic cells in peripheral blood after achieving complete remission, or bone marrow blast count > 5% (excluding other causes such as bone marrow reconstitution post-consolidation chemotherapy), or the presence of extramedullary leukemic cell infiltration.
2. . Ineligible for bone marrow transplantation, or have undergone bone marrow transplantation but failed to achieve long-term remission.

4. Expression of both CLL-1 and CD70 targets is confirmed as positive by flow cytometry.

5. Patients must have good major organ function:

1. . Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤ 34.2 μmol/L.
2. . Kidney function: Creatinine clearance rate (Cockcroft-Gault method) ≥ 60 mL/min.
3. . Lung function: Oxygen saturation ≥ 95%, with no active pulmonary infection.
4. . Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; no significant pericardial effusion, and no clinically significant ECG abnormalities.

6. Women of childbearing age must have a negative urine/blood pregnancy test during screening and agree to use contraceptive measures for at least 1 year after infusion. Male subjects with reproductive capacity must agree to use effective barrier contraception for at least 1 year after infusion.

7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-3. 8. Expected life expectancy greater than 3 months. 9. The patient is willing to cooperate with the collection of peripheral blood mononuclear cells, medical examinations, and regular follow-up visits.

Exclusion Criteria:

The patient will be excluded if meeting any of the following criteria:

1. Women who are pregnant or breastfeeding.
2. Presence of uncontrolled fungal, bacterial, treponemal (e.g., syphilis), viral, or other infections.
3. Active hepatitis B (Hepatitis B virus DNA > 500 IU/mL) or a positive Hepatitis C virus RNA (HCV-RNA) test.
4. Human Immunodeficiency Virus (HIV) infection, or syphilis infection.
5. Previously received any form of gene therapy.
6. The patient has an allergic constitution or is allergic to macromolecular biologics such as antibodies or cytokines.
7. History of clinically significant central nervous system diseases, such as: epilepsy, hemiparesis, aphasia, stroke, severe brain trauma, dementia, Parkinson's disease, cerebellar diseases, or organic brain syndromes.
8. Uncontrolled psychiatric illness.
9. A history of drug abuse/addiction.
10. Use of prohibited medications:

(1). Hormones: Use of corticosteroids (prednisone ≥ 2 mg/kg or equivalent > 20 mg/day) within 2 weeks prior to cell collection. Recent or ongoing use of inhaled, topical, or non-absorbable steroids is not an exclusion criterion.

(2). Radiotherapy/Chemotherapy:Receipt of radiotherapy or salvage chemotherapy for the study disease within 3 weeks prior to cell collection.

(3). Use of immunosuppressive agents within 4 weeks prior to cell collection. (4). Participation in another clinical trial or receipt of a major non-diagnostic surgical procedure within 4 weeks prior to cell collection.

(5). Use of alemtuzumab within 6 months, or cladribine/clofarabine within 3 months, prior to cell collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  The overall response rate (ORR) includes both complete response (CR) and partial response (PR), and uses the Clopper-Pearson method to calculate the two-sided 95% confidence interval.

IPD SHARING:
Plan to Share IPD: No